CLINICAL TRIAL: NCT04069572
Title: Patterned Multichannel Vibratory Coordinated Reset (VCR) Stimulation for the Treatment of Chronic Pain
Brief Title: Vibratory Stimulation for the Treatment of Chronic Pain
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: New investigational devices are currently under development.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Hah, Assistant Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 52019
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain; Pelvic Pain; Functional Abdominal Pain Syndrome; Low Back Pain; Migraine
MeSH Terms: conditions — Chronic Pain; Pelvic Pain; Low Back Pain; Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vibrotactile Stimulation (Experimental)
  Interventions: Device: Vibrotactile Stimulation
- Sham Stimulation (Sham Comparator)
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Vibrotactile Stimulation — Application of VCR stimulation to the belly and back of patients with pelvic pain, functional abdominal pain, or low back pain or to the temporal region for patients with migraine.
  Arms: Vibrotactile Stimulation
Device: Sham Stimulation — Low-frequency sham of VCR stimulation
  Arms: Sham Stimulation

SUMMARY:
The purpose of this study is to perform a first in man study with VCR stimulation of the belly and back for patients with chronic pain conditions including pelvic pain, functional abdominal pain, or low back pain. This study will also examine VCR stimulation of the temporal region for patients with migraine with or without aura. Additional goals of the study will be to determine the safety, tolerability, and acceptability of VCR stimulation for the treatment of these pain conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old.
* Diagnosis of either chronic pelvic pain, functional abdominal pain, axial low back pain, or migraine with or without aura of at least 3 months duration.
* English speaking
* Ability and willingness to complete questionnaires and in-person assessments
* Current average daily pain score of greater than or equal to 4 on the Numeric Rating Scale of Pain (0-10 scale)
* For patients with migraine diagnosis they must report at least 2 headaches in the baseline headache diary in the 30 days preceding randomization.

Exclusion Criteria:

* Any conditions causing inability to complete assessments (education, cognitive ability, mental status, medical status)
* Any significant psychiatric problems, including acute confusional state (delirium), ongoing psychosis, or clinically significant depression
* Any suicidality as assessed by answer of greater than 0 on question 9 the PHQ-9 assessing suicidal thoughts.
* Any current illicit drug or alcohol abuse.
* Any history of recurrent or unprovoked seizures.
* Participation in another drug, device, or biologics trial concurrently or within the preceding 30 days.
* Pregnancy, breast-feeding or lack of reliable contraception
* Changes in pain medications in the previous 4 weeks
* Implanted electrical stimulation device.
* Skin infection over stimulation sites.
* Any pain interventions in the preceding 6 weeks (epidural steroid injection, sympathetic block, peripheral nerve block, lumbar medial branch blocks) Any botulinum toxin injection in the previous 3 months
* For patients with migraine diagnosis additional exclusion criteria include receipt of preventive anti-migraine treatment in the past 3 months, failure on greater than or equal to 3 well-conducted preventive drug trials, concurrent medication overuse headache diagnosis, and concurrent frequent/chronic tension type headache.

  4. Frequent/chronic tension type headache

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Treatment Responder | 30 days
  Proportion of subjects in the treatment vs. placebo groups that are responders with greater than or equal to 50% reductions in average pain (in the primary pain area) comparing the average pain score from the 7-day baseline diary pre-treatment to the average scores based on 7-day diaries at the end of the primary outcome interval
Change in Opioid Use | 30 days
  Change in opioid use in daily oral morphine equivalents from the average 7-day baseline use to the post-treatment use in the 7 days at the end of the primary outcome interval.

SECONDARY OUTCOMES:
Adverse Events | 60 days
  The proportion of adverse events occurring in the treatment vs. placebo groups
Secondary Treatment Response After Crossover | 60 days
  The proportion of subjects in the treatment vs. placebo groups that are responders at the end of 60 days comparing the average pain score from the 7- day baseline diary pre-treatment to the reported pain score at the end of the 60 day interval.
Change in monthly migraine days | 30 days
  For patients with migraine, change in monthly migraine days between the 30 days before randomization and the end of the primary outcome interval.
Treatment Engagement | 30 days
  Treatment engagement is defined as participation in >50% of home treatment sessions.
Treatment Initiation | 30 days
  Treatment initiation is defined as participation in at least 1 home treatment session. session.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Hah, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Neuroscience Health Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No